CLINICAL TRIAL: NCT01812746
Title: An Open Label, Multicenter, Phase 2 Study to Determine the Safety and Efficacy of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension), Administered to Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase 2 Study to Determine the Safety and Efficacy of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension), Administered to Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIND-014-004
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: CRPC; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- BIND-014 (Experimental)
  Interventions: Drug: BIND-014

INTERVENTIONS:
Drug: BIND-014

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety BIND-014 in patients with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Metastatic disease progressing despite castrate levels of testosterone
* Prostate cancer progression documented by PSA
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL
* Previous anti-androgen therapy and progression after withdrawal
* ECOG performance status of 0 to 1
* Adequate organ function
* Prior radiation therapy allowed to < 25% of the bone marrow
* Prior hormonal therapy is allowed
* Patient compliance and geographic proximity that allow adequate follow-up.
* Patients with reproductive potential must use contraceptive methods
* Signed informed consent from patient

Exclusion Criteria:

* Active infection
* Any chronic medical condition requiring a high doses of corticosteroid
* Pathological finding consistent with small cell carcinoma of the prostate
* Brain metastasis
* Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
* Radiation therapy for treatment of the primary tumor within 6 weeks
* Radionuclide therapy for treatment of metastatic CRPC
* Prior systemic treatment with an azole drug
* Prior flutamide treatment within 4 weeks
* Prior bicalutamide or nilutamide within 6 weeks
* Congenital long QT syndrome, congestive heart failure, or bradyarrhythmia
* Administration of an investigational therapeutic within 2 weeks
* Second primary malignancy
* Presence of clinically detectable third-space fluid collections
* History of severe hypersensitivity reaction to polysorbate 80
* Peripheral neuropathy at study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of BIND-014 as measured by radiographic progression-free survival (rPFS) in patients with chemotherapy-naïve metastatic CRPC | Patients will be followed for the duration of treatment, an expected average of 24 weeks
  Number of patients with a progression-free survival of 6 months

SECONDARY OUTCOMES:
To assess the safety and tolerability of BIND-014 | Patients will be followed for the duration of treatment, an expected average of 24 weeks
  Number of patients who experience adverse events

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Investigative Site #16, Los Angeles, California
  - Investigative Site #14, San Francisco, California
  - Investigative Site #17, Fort Meyers, Florida
  - Investigational Site #12, Ann Arbor, Michigan
  - Investigational Site #11, New York, New York
  - Investigational Site #15, Chapel Hill, North Carolina
  - Investigational Site #13, Cleveland, Ohio
  - Investigational Site #18, Nashville, Tennessee

REFERENCES:
- [Background] Hrkach J, Von Hoff D, Mukkaram Ali M, Andrianova E, Auer J, Campbell T, De Witt D, Figa M, Figueiredo M, Horhota A, Low S, McDonnell K, Peeke E, Retnarajan B, Sabnis A, Schnipper E, Song JJ, Song YH, Summa J, Tompsett D, Troiano G, Van Geen Hoven T, Wright J, LoRusso P, Kantoff PW, Bander NH, Sweeney C, Farokhzad OC, Langer R, Zale S. Preclinical development and clinical translation of a PSMA-targeted docetaxel nanoparticle with a differentiated pharmacological profile. Sci Transl Med. 2012 Apr 4;4(128):128ra39. doi: 10.1126/scitranslmed.3003651. PMID 22491949
- [Derived] Autio KA, Dreicer R, Anderson J, Garcia JA, Alva A, Hart LL, Milowsky MI, Posadas EM, Ryan CJ, Graf RP, Dittamore R, Schreiber NA, Summa JM, Youssoufian H, Morris MJ, Scher HI. Safety and Efficacy of BIND-014, a Docetaxel Nanoparticle Targeting Prostate-Specific Membrane Antigen for Patients With Metastatic Castration-Resistant Prostate Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Oct 1;4(10):1344-1351. doi: 10.1001/jamaoncol.2018.2168. PMID 29978216